CLINICAL TRIAL: NCT01097538
Title: Total Body Recumbent Stepper Training in Progressive MS: An Alternative Training Therapy for Patients With Impaired Mobility
Brief Title: Study of Alternative Exercise Therapies for Progressive Multiple Sclerosis (MS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hicks, Audrey, Ph.D. (Individual)
Responsible Party: Audrey Hicks, PhD. (Professor), McMaster University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Hicks -MS exercise
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Multiple Sclerosis
Keywords: exercise; rehabilitation; progressive multiple sclerosis; functional ability; fatigue; quality of life
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Multiple Sclerosis, Chronic Progressive; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Body-weight supported treadmill training (Active Comparator): Supported treadmill walking
  Interventions: Other: Body-weight supported treadmill training
- Total body recumbent stepper training (Experimental): Recumbent stepper exercise training
  Interventions: Other: Total body recumbent stepper training

INTERVENTIONS:
Other: Body-weight supported treadmill training — Patients will undergo training using the Woodway Loco-system which consists of a treadmill with an overhead pulley system connected to a support harness. BWSTT allows patients with limited mobility to safely walk upright on a treadmill with a portion of their body weight counter balanced. Three trainers will be required to assist with the BWSTT program. Two trainers will be positioned at the lower limbs to manually guide the participant through a proper gait motion and provided lower limb control. A third trainer will stand behind the participant to provide trunk support and assist with weight shifting.
  Arms: Body-weight supported treadmill training
Other: Total body recumbent stepper training — Patients will train using the Nustep T4 (TRS 4000) which is a recumbent cross trainer that provides a full body workout in a seated position. The Nustep trainer allows patients to achieve a natural stepping motion against graded loads with bilateral reciprocal movement of the arms. Recumbent training is safe and easily accessible for patients of all ability levels with a swivel chair to aid in patient transfers. Foot straps, leg stabilizers and hand stabilizers may be used for added control and proper body alignment.
  Arms: Total body recumbent stepper training

SUMMARY:
This project will evaluate a new therapy for patients with a severe form of MS known as progressive MS. These patients are severely limited in their ability to walk and function in everyday life. The exercise therapy we are proposing is a recumbent cross trainer which allows patients to be seated and move their arms and legs at the same time against resistive foot pedals and arm levers. The recumbent cross trainer is safe and easy to use for people with disabilities and is more cost-effective compared with other rehabilitation equipment. Before the recumbent trainer can become part of mainstream MS therapy, it is important to determine if it is as effective as other exercise therapies in improving functional performance and quality of life. In this study we will compare the effects of the recumbent cross training with supported treadmill walking on functional and psychological outcomes. Further, since this is a new therapy for progressive MS patients, we also want to determine if it is safe and enjoyable to use.

We hypothesize that recumbent stepper training will be safe and well-tolerated by progressive MS patients. Both training interventions will be beneficial in improving walking function and psychosocial outcomes. Recumbent stepper straining will likely have greater effects on upper extremity function, while supported treadmill walking will have greater effects on lower extremity function.

DETAILED DESCRIPTION:
We are proposing to evaluate the clinical utility and efficacy of a new therapeutic exercise modality for patients with progressive MS with severe functional impairments.

Progressive MS patients have limited treatment options and reach higher disability levels at a faster rate than relapsing remitting MS patients. Consequently, finding solutions to maintain function and improve quality of life of patients with progressive MS is essential.

A traditional training modality for patients with limited mobility is body-weight supported treadmill training (BWSTT). Our preliminary results support the efficacy of BWSTT in progressive MS patients; however, the financial burden and labour-intensive nature of BWSTT does not make it a viable option for most settings. For the aforementioned reasons, we are proposing total body recumbent stepper training (TBRST) as an alternative therapy for progressive MS patients with mobility impairments. TBRST is advantageous over BWSTT in that it has low set-up and maintenance costs, is easily used by patients with limited mobility and requires minimal assistance to operate. TBRST has the potential to become part of conventional MS treatment programs and could easily be incorporated into home and community settings. The primary aim of this investigation is to establish safety and satisfaction with TBRST in progressive MS patients. Second, we plan to determine if TBRST is as effective as a BWSTT as a therapeutic modality.

Twenty patients with progressive MS (primary and secondary) of high disability level (EDSS 6.0-8.0) will be recruited to participate in this study. Both primary and secondary MS patients will be included due to similarities in disease progression and a lack of available alternative treatments for this population. Patients will be randomized to either the TBRST or BWSTT intervention; there will be 10 patients in each group. Patients in the TBRST program will train using the Nustep (TRS 4000) recumbent cross trainer. The recumbent cross trainer allows patients to move their legs in a natural stepping motion with bilateral reciprocal movement of the arms from a seated position. Foot straps, leg stabilizers and hand stabilizers may be used for added control and proper body alignment when necessary. Patients in the BWSTT group will exercise using the Woodway Loco-system which allows a portion of the patient's body-weight to be off-loaded by an overhead pulley system. Treadmill therapists will guide the patients' legs through a proper gait motion and assist with lower limb control.

Participants in both interventions will complete three weekly exercise sessions of 30min, for the duration of 12 weeks. Perceived exertion will be used as an indicator of exercise intensity and will guide program progression. Both intervention groups will maintain a perceived exertion of 5-7 on the Borg CR10 Scale throughout the exercise program. All patients will be evaluated at baseline and following 12 weeks on a variety of outcome measures. Primary outcome measures will be safety and satisfaction with TBRST. Secondary outcomes will be functional ability using the EDSS and MSFC, quality of life using the MSQOL-54, fatigue using the MFIS and MS self-efficacy using the MSSE. The proposed research will take place over one year with enrolment and intervention programs commencing in a graded manner.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent
* Males or non-pregnant females, 18-60 years of age (inclusive)
* Clinically definite PPMS as per the diagnostic criteria of Thompson et al OR clinically definite SPMS as per the diagnostic criteria of McDonald et al for RRMS with slow gradual progression observed over 6 months, not due to deterioration from attacks alone
* Absence of a relapse in the previous 6 months
* Expanded disability status score 6.0-8.0 (constant assistance required)
* Body weight <90kg (due to support limitations of treadmill)
* Approval from physician to participate in the exercise program
* Ability to tolerate upright locomotion of the body weight supported treadmill
* Ability to visit the different sites required for the study
* Ability to commit to 3 weekly training sessions during specified training times for the duration of 12 weeks
* Ability to follow training instructions

Exclusion Criteria:

* Any disability acquired from trauma or another illness that could interfere with evaluation of disability due to MS
* Any other serious medical condition that might impair the subject's ability to walk on a treadmill and/or participate in aerobic exercise (including but not limited to: documented heart disease or unstable angina, uncontrolled cardiac dysrhythmia, chronic obstructive lung disease, recent non-traumatic fracture, osteoporosis and severe skin ulcerations)
* Female patients who do not agree to use effective contraceptive method(s) during the study
* Current use or use within the last 2 months of any on- or off-label disease-modifying therapy including IFN-β, glatiramer acetate, IV steroids, mitoxantrone, azathioprine, and cyclophosphamide
* Previous experience with recumbent stepper training or supported treadmill training

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety | baseline, 12 weeks (end of trial)
  Adverse effects will be monitored at each training session. Therapists will record patient experiences of muscle and joint pain, physical discomfort, excessive fatigue, overheating, chest pain, dizziness/nausea and any other adverse effects experience by the patients. If symptoms become severe patients will be asked to discontinue training and consult their physician immediately.

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) -neurologic function | baseline, 12 weeks (end)
  The EDSS provides a measure of physical function specifically in MS patients and is scored from 0-10. This will be assessed by a train neurologist.
Multiple Sclerosis Functional Composite (MSFC)-functional ability | baseline, 12 weeks (end)
  The MSFC assesses functional ability with three scales: the 25ft walk (leg strength and ambulation), the 9-hole peg test (arm strength and coordination) and the Paced Auditory Serial Addition Test (PASAT; cognition). Scores on all three measures are combined to produce a composite Z-score.
Modified Fatigue Impact Scale (MFIS) -fatigue | baseline, 12 weeks (end)
  The MFIS is a 21-item self-report questionnaire that evaluates fatigue overall fatigue, as well as within three categories: physical (pMFIS); cognitive (cMFIS); and psychosocial (psMFIS), over the previous 4 weeks. Scores range from 0-4 on each item with a maximum total score of 84, where higher scores indicate greater fatigue levels.
Multiple Sclerosis Quality of Life-54 -quality of life questionnaire | baseline, 12 weeks (end)
  The MSQOL-54 is an MS-specific measure of QOL that consists of 54 items divided into 12 multi-item scales, 2 single-item scales, and 2 composite scores (physical and mental health).
Multiple Sclerosis Self-Efficacy Scale (MSSE) -ability to manage MS symptoms | baseline, 12 weeks (end)
  The MSSE is an 18-item questionnaire which evaluates self-efficacy on two multi-item subscales: function and control. Each subscale ranges from 10 (very uncertain) to 100 (very certain) on how certain the individual is in their function or control of their MS symptoms.
Participant Satisfaction with Equipment | once -following 5 full exercise sessions
  In order to assess satisfaction with equipment, patients will be asked a series of questions concerning the accessibility, perceived benefit, enjoyment and after-effects of using both equipment modalities. This questionnaire is composed of a series of scales compiled from a number of sources including the Brief Pain Inventory, the Feeling Scale and the Exercise Feeling Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Hicks, PhD, Principal Investigator — McMaster University; Lara Pilutti, Principal Investigator — McMaster University
Locations (1):
- Centre for Health Promotion and Rehabilitation, McMaster University, Hamilton, Ontario, Canada